CLINICAL TRIAL: NCT02254642
Title: Protective Effects of Ischemic Preconditioning on Cardiac, Renal, Pulmonary and Muscular Functions After Aortic Clamping
Brief Title: Effects of Ischemic Preconditioning After Aortic Clamping
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5831
Record Dates: First submitted 2014-06-26; First posted 2014-10-02 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Vascular Surgery; Ischemia-reperfusion; Ischemia Preconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic preconditioning arm (Experimental): Patients will have the ischemic preconditioning protocol 1 hour before the aortic clamping.
  Interventions: Procedure: Ischemic preconditioning during aortic clamping
- Control patients (Other): Usual surgery assigned to control patients
  Interventions: Procedure: Procedure/Surgery: usual surgery

INTERVENTIONS:
Procedure: Ischemic preconditioning during aortic clamping — Ischemic preconditioning during aortic clamping
  Arms: Ischemic preconditioning arm
Procedure: Procedure/Surgery: usual surgery — Procedure/Surgery: usual surgery
  Arms: Control patients

SUMMARY:
Open surgery for aneurysmal aortic disease can lead to cardiac, renal, pulmonary or muscular complications, essentially due to the aortic clamping. Ischemic preconditioning can be useful in order to decrease these complications. The investigators would like to use an ischemic preconditioning protocol during open surgery of aortic aneurysm in order to decrease these complications.

ELIGIBILITY:
Inclusion criteria:

* Patients with an aortic aneurysm requiring open surgery (with no possibility of endovascular surgery)
* Patients who received clear information, with signed consent
* Patients 18 to 85 years

Exclusion criteria:

* Patients under guardianship
* No possibility to give the patients clear information (comprehension difficulties, emergency surgery)
* Pregnancy, lactation
* Hemodialysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Myocardial damage measured by troponin level > 0.4 microgr/L (day 1) | Day 1
  Myocardial damage measured by Troponin I level > 0.4 microg/L

SECONDARY OUTCOMES:
Renal damage | Day 0, day 1, day 3 or day 5.
  Renal damage measured with Post-operative Creatinin clearance < 50% of Pre-operative creatinin clearance
Muscle weakness | Day 0, day 1, day 3 or day 5
  Muscle weakness measured by Creatine phospho Kinase > 200 UI/L
Myocardial damage measured by troponin level > 0.4 microgr/L | Day 0, 3, or 5

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lejay, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Service de Chirurgie Vasculaire, CH Jean Minjoz, Besançon
  - Service de Chirurgie Vasculaire, CHU le Bocage, Dijon
  - Service de Chirurgie vasculaire et transplantation rénale, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Chirurgie Vasculaire, Hôpitaux Privés de Metz, Site de Mercy, Vantoux

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250